CLINICAL TRIAL: NCT02977962
Title: Treatment of Anxiety in Late Adolescents With Autism
Acronym: TALAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of South Florida (Other)
Collaborators: Johns Hopkins All Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: USF-ACH 001
Record Dates: First submitted 2016-11-28; First posted 2016-11-30 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Cognitive Behavioral Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-Behavior Therapy (Experimental): This consists of 16 weekly sessions up to 90 minutes each that helps the participant learn to cope with anxiety by facing fears, thinking more logically, and calming oneself.
  Interventions: Behavioral: Cognitive-Behavior Therapy
- Treatment as Usual (Placebo Comparator): Participants randomized to this condition will wait for a period of 16 weeks before receiving treatment in the context of the study. During this time, youth may receive psychotherapy and/or initiate or change current psychiatric medication (if applicable).
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Cognitive-Behavior Therapy — This therapy has been designed for adolescents with high functioning ASD and involves 16 weekly session where the participant learns coping skills related to addressing anxiety (e.g., exposure therapy, cognitive therapy, social skills training).
  Other Names: CBT
  Arms: Cognitive-Behavior Therapy
Other: Treatment as Usual — Those who choose to participate will be enrolled in the 16 week study. They will required to attend 3 assessments - pre-treatment (week 0), mid-treatment (week 8), and post-treatment (week 16). Those in this group will not receive the Cognitive-Behavior Therapy, and instead will undergo therapy for their anxiety as they usually would, whether by using medication or working with a therapist.
  Arms: Treatment as Usual

SUMMARY:
Autism spectrum disorders (ASD) affect approximately 1.1% of late adolescents and young adults, making it one of the most common neurodevelopmental disorders. Comorbid anxiety disorders affect many higher-functioning adolescents and young adults with ASD, causing substantial distress and impairment over and above that caused by an ASD diagnosis alone. While cognitive-behavioral therapy (CBT) is a first-line treatment for anxiety disorders among typically developing late adolescents, and work by the investigative team supports its utility in children with ASD and comorbid anxiety, very few evidence-based treatment approaches exist for late adolescents with ASD and comorbid anxiety. Accordingly, the investigators are proposing to develop a CBT protocol for clinical anxiety that is personalized to the unique clinical characteristics of late adolescents (ages 16-21 years) with ASD namely, the Treatment of Anxiety in Late Adolescents with Autism (TALAA).

DETAILED DESCRIPTION:
Autism spectrum disorders (ASD) affect approximately 1.1% of late adolescents and young adults, making it one of the most common neurodevelopmental disorders. Comorbid anxiety disorders affect many higher-functioning adolescents and young adults with ASD, causing substantial distress and impairment over and above that caused by an ASD diagnosis alone. While cognitive-behavioral therapy (CBT) is a first-line treatment for anxiety disorders among typically developing late adolescents, and work by the investigative team supports its utility in children with ASD and comorbid anxiety, very few evidence-based treatment approaches exist for late adolescents with ASD and comorbid anxiety. Accordingly, the investigators are proposing to develop a CBT protocol for clinical anxiety that is personalized to the unique clinical characteristics of late adolescents (ages 16-21 years) with ASD namely, the Treatment of Anxiety in Late Adolescents with Autism (TALAA). Initial TALAA development efforts will focus on adapting relevant treatment elements from an efficacious CBT program for early adolescents with ASD and comorbid anxiety to the characteristics and clinical needs of the age group. Developmentally appropriate, novel treatment components will be added, including those focusing on fostering successful transitions to adulthood (e.g., work readiness). In response to the NIH Roadmap Initiative, attention will be paid to protocol adaptability with varying clinical presentations. Measures of treatment integrity and competence will be developed. Thereafter, protocol and measure development will be refined through our experiences treating 8 young adults (ages 16-21 years) with ASD and comorbid anxiety disorder(s) as well as through clinician, patient, and expert feedback. The feasibility of implementing TALAA will then be examined in the context of a pilot study incorporating all the features of the planned future efficacy trial comparing TALAA to treatment as usual, but with a limited sample size (N=44).

ELIGIBILITY:
Inclusion Criteria:

* Outpatient males and females with ASD between the ages 16-21 years at consent/assent.
* The individual meets criteria for ASD.
* The individual meets criteria for clinically significant anxiety symptoms.
* Meets criteria for a diagnosis of one of the following anxiety disorders: separation anxiety disorder (SAD), specific phobia, panic disorder (PD), generalized anxiety disorder (GAD), social phobia (SP), or obsessive compulsive disorder (OCD) and has a minimum score of 14 on the Hamilton Anxiety Scale.
* Person has a Full Scale IQ approximation > 70 as assessed by the Wechsler Abbreviated Scale for Intelligence-II two or four sub-test form.

Exclusion Criteria:

* Receiving concurrent psychotherapy focused on anxiety.
* Initiation of an antidepressant medication within 12 weeks before study enrollment or an antipsychotic medication 6 weeks before study enrollment or the child has changed the dose of an established medication within 8 weeks before study enrollment (4 weeks for antipsychotic) or during psychotherapy (unless the dose is lowered because of side effects).
* (a) Current clinically significant suicidality or (b) individuals who have engaged in suicidal behaviors within 6 months will be excluded and referred for appropriate clinical intervention.
* Lifetime bipolar disorder, schizophrenia or schizoaffective disorder, or substance abuse in past 6 months.

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-01; Primary Completion 2021-04 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in anxiety severity on the Hamilton Anxiety Scale after 16 weeks of treatment. | After 16 weeks of treatment
  This measure is administered by a clinician and assesses anxiety with scores between 0-30. Higher ratings correspond to more severe anxiety symptoms.

SECONDARY OUTCOMES:
Change from Baseline in anxiety severity on the Clinical Global Impressions Scale after 16 weeks of treatment. | After 16 weeks of treatment
  This measure is completed by the clinician and assesses the severity of anxiety on a 7 point scale (0-6; higher scores correspond to worse anxiety).

CONTACTS AND LOCATIONS:
Overall Officials: Adam Lewin, Ph.D., Principal Investigator — University of South Florida
Locations (1):
- Rothman Center for Neuropsychiatry, University of South Florida, St. Petersburg, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elliott SJ, Marshall D, Morley K, Uphoff E, Kumar M, Meader N. Behavioural and cognitive behavioural therapy for obsessive compulsive disorder (OCD) in individuals with autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2021 Sep 3;9(9):CD013173. doi: 10.1002/14651858.CD013173.pub2. PMID 34693989